CLINICAL TRIAL: NCT01478581
Title: A Multicenter Phase 2 Study of the Bruton's Tyrosine Kinase (Btk) Inhibitor, PCI-32765, in Subjects With Relapsed or Relapsed and Refractory Multiple Myeloma
Brief Title: Study of the Bruton's Tyrosine Kinase Inhibitor in Subjects With Relapsed or Relapsed and Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-1111-CA; PCI-32765 (Other: Sponsor)
Record Dates: First submitted 2011-11-18; First posted 2011-11-23 (Estimated); Results first posted 2018-06-26 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2019-10

CONDITIONS: Multiple Myeloma
Keywords: PCI-32765; Multiple Myeloma; Relapsed Refractory Multiple Myeloma; Bruton's Tyrosine Kinase
MeSH Terms: conditions — Multiple Myeloma | interventions — ibrutinib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): PCI-32765 420 mg per day
  Interventions: Drug: PCI-32765
- Cohort 2 (Experimental): PCI-32765 560 mg per day, 40 mg dexamethasone (oral) once per week
  Interventions: Drug: PCI-32765; Drug: Dexamethasone
- Cohort 3 (Experimental): PCI-32765 840 mg per day
  Interventions: Drug: PCI-32765
- Cohort 4 (Experimental): PCI-32765 840 mg per day, 40 mg dexamethasone (oral) once per week
  Interventions: Drug: PCI-32765; Drug: Dexamethasone

INTERVENTIONS:
Drug: PCI-32765
  Other Names: Ibrutinib
Drug: Dexamethasone
  Arms: Cohort 2; Cohort 4

SUMMARY:
The primary objective of this study is to determine the efficacy of PCI-32765, both as a single agent and in combination with dexamethasone, in subjects with relapsed or relapsed and refractory Multiple Myeloma (MM)

DETAILED DESCRIPTION:
Bruton's tyrosine kinase (Btk) is an enzyme that is present in hematopoietic cells other than T cells and is necessary for downstream signal transduction from various hematopoietic receptors including the B cell receptor as well as some Fc, chemokine, and adhesion receptors, and is crucial for both B cell development and osteoclastogenesis. Although down-regulated in normal plasma cells, Btk is highly expressed in the malignant cells from many myeloma patients and some cell lines. PCI 32765 is a potent and specific inhibitor of Btk currently in Phase 2 clinical trials. The current study is designed and intended to determine the effects of PCI-32765 in subjects with MM.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of symptomatic MM with measurable disease, defined here as having at least one of the following:

  1. Serum monoclonal protein (M-protein) ≥0.5 g/dL as determined by serum protein electrophoresis (SPEP)
  2. Urine M-protein ≥200 mg/24 hrs
  3. Serum free light chain (FLC) assay: involved FLC level ≥10 mg/dL (≥100 mg/L) provided serum FLC ratio is abnormal
* Relapsed or relapsed and refractory MM after receiving at least 2 but no more than 5 previous lines of therapy, 1 of which must be an immunomodulator.
* Refractory myeloma (to most recent treatment) is defined as disease that is nonresponsive while on treatment or progressive disease within 60 days after the completion of preceding treatment. Nonresponsive disease is defined as either failure to achieve minimal response or development of progressive disease while on therapy.
* Men and women ≥18 years of age.
* ECOG performance status of ≤ 1.

Exclusion Criteria:

* Subject must not have primary refractory disease defined as disease that is nonresponsive in subjects who have never achieved a minor response (MR) or better with any therapy.
* Polyneuropathy, organomegaly, endocrinopathy, M-protein, and skin changes (POEMS) syndrome, osteosclerotic myeloma, or Crow-Fukase syndrome.
* Plasma cell leukemia.
* Primary amyloidosis.
* Certain exclusions on prior therapy.
* ANC <0.75 x 10^9/L independent of growth factor support.
* Platelets <50 x 10^9/L) independent of transfusion support.
* AST or ALT ≥3.0 x upper limit of normal (ULN).
* Total bilirubin >2.5 x ULN, unless due to Gilbert's syndrome.
* Creatinine >2.5 mg/dL.
* Unable to swallow capsules or disease significantly affecting gastrointestinal function.
* Requires anti-coagulation with warfarin or a vitamin K antagonist. Requires treatment with strong CYP3A4/5 inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - SITE-13, La Jolla, California
  - SITE-5, Baltimore, Maryland
  - SITE-4, Boston, Massachusetts
  - SITE-8, Ann Arbor, Michigan
  - SITE-2, St Louis, Missouri
  - SITE-6, Hackensack, New Jersey
  - SITE-10, New York, New York
  - SITE-3, New York, New York
  - SITE-1, Nashville, Tennessee
  - SITE-11, Dallas, Texas
  - SITE-9, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Simon 2-stage design . Stage 1 -13 subjects enrolled in cohort 1. For cohort 2,3, and 4, up to 18 subjects were enrolled in Stage 1. Cohort 4 was selected for expansion for enrollment of 43 subjects in Stage 2.
Groups:
- PCI-32765 420 mg Per Day: PCI-32765 420 mg per day
  PCI-32765
- PCI-32765 560 mg Per Day, 40 mg Dexamethasone: PCI-32765 560 mg per day, 40 mg dexamethasone (oral) once per week
  PCI-32765
  Dexamethasone
- PCI-32765 840 mg Per Day: PCI-32765 840 mg per day
  PCI-32765
- PCI-32765 840 mg Per Day, 40 mg Dexamethasone: PCI-32765 840 mg per day, 40 mg dexamethasone (oral) once per week
  PCI-32765
  Dexamethasone
Period: Overall Study
Arm/Group | PCI-32765 420 mg Per Day | PCI-32765 560 mg Per Day, 40 mg Dexamethasone | PCI-32765 840 mg Per Day | PCI-32765 840 mg Per Day, 40 mg Dexamethasone
Started | 13 | 18 | 18 | 43 (Simon 2-stage design - cohort 4 expansion per stage 1 data (≥3 Clinical Benefit Responders observed)
Completed | 13 | 18 | 18 | 43
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: PCI-32765 420 mg per day
  PCI-32765
- Cohort 2: PCI-32765 560 mg per day, 40 mg dexamethasone (oral) once per week
  PCI-32765
  Dexamethasone
- Cohort 3: PCI-32765 840 mg per day
  PCI-32765
- Cohort 4: PCI-32765 840 mg per day, 40 mg dexamethasone (oral) once per week
  PCI-32765
  Dexamethasone
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 13 | 18 | 18 | 43 | 92
Age, Continuous [Median (Standard Deviation); unit: years] | 62.0 (7.57) | 65.5 (8.44) | 65.5 (7.52) | 65.0 (7.40) | 65.0 (7.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 5 | 17 | 36
  Male | 8 | 9 | 13 | 26 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 6 | 7
  Not Hispanic or Latino | 13 | 18 | 17 | 34 | 82
  Unknown or Not Reported | 0 | 0 | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — We have 5 patients with Race reported as "Other". For these 5 patients we reported the race data under "Unknown or Not Reported" as no "Other" category available in this database.
  Participants
    Other Race: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Other Race: Asian | 0 | 0 | 1 | 0 | 1
    Other Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Other Race: Black or African American | 2 | 6 | 4 | 6 | 18
    Other Race: White | 10 | 12 | 12 | 33 | 67
    Other Race: More than one race | 0 | 0 | 1 | 0 | 1
    Other Race: Unknown or Not Reported | 1 | 0 | 0 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 13 | 18 | 18 | 43 | 92

OUTCOME MEASURES:

1. Primary Outcome: The Clinical Benefit Response (CBR)
Description: The clinical benefit response (CBR) rate, defined as the proportion of subjects who achieved stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), or minimal response (MR) as assessed by the modified International Myeloma Working Group (IMWG) response criteria
Time Frame: From the date of first study treatment until disease progression per IMWG, up to 60 months
Population: All treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 13 | 18 | 18 | 43
Participants | 1 | 1 | 0 | 12

2. Secondary Outcome: To Evaluate the Efficacy of PCI-32765 by Assessing ORR
Description: The objective response rate, defined as the proportion of subjects who achieved stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR), as assessed by the modified International Myeloma Working Group (IMWG) response criteria.
Time Frame: From the date of first study treatment until disease progression per IMWG, up to 60 months
Population: All treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 13 | 18 | 18 | 43
Participants | 0 | 1 | 0 | 2

3. Secondary Outcome: Pharmacokinetics (PK). (Assessed by Sampling and Testing for Drug and Metabolite Levels at Designated Time Points). Mean Maximum Observed Plasma Concentration (Cmax)
Description: Ibrutinib and PCI-45227 concentrations were measurable following once-daily dosing of ibrutinib in subjects with MM. The following time-points were included: 0hr, 1hr, 2hr, 7hr, 24hr post-dose. Maximum observed plasma concentration of ibrutinib during the dosing interval on Day 8.
Time Frame: Procedure was performed up to 60 weeks.
Population: All subjects who received at least one dose of study treatment and had evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 13 | 16 | 18 | 43
ng/mL | 157 (126) | 103 (96.7) | 219 (159) | 166 (200)

4. Secondary Outcome: Pharmacokinetics (PK) (Assessed by Sampling and Testing for Drug and Metabolite Levels at Designated Time Points). Mean Time to Maximum Observed Plasma Concentration (Tmax).
Description: Ibrutinib and PCI-45227 concentrations were measurable following once-daily dosing of ibrutinib in subjects with MM. The following time-points were included: 0hr, 1hr, 2hr, 7hr, 24hr post-dose. Time to corresponding maximum observed plasma concentration of ibrutinib during the dosing interval on Day 8.
Time Frame: Procedure was performed up to 60 weeks.
Population: All subjects who received at least one dose of study treatment and had evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 13 | 16 | 18 | 43
hours | 2.73 (1.99) | 2.32 (1.72) | 1.95 (0.944) | 2.25 (1.18)

5. Secondary Outcome: Pharmacokinetics (PK) (Assessed by Sampling and Testing for Drug and Metabolite Levels at Designated Time Points). Mean Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours (AUC0-24h).
Description: Ibrutinib and PCI-45227 concentrations were measurable following once-daily dosing of ibrutinib in subjects with MM. The following time-points were included: 0hr, 1hr, 2hr, 7hr, 24hr post-dose. Ibrutinib AUC0-24h calculated using linear trapezoidal summation after dosing from time 0 to 24 hours on Day 8.
Time Frame: Procedure was performed up to 60 weeks.
Population: All subjects who received at least one dose of study treatment and had evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: h∙ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 13 | 16 | 18 | 43
h∙ng/mL | 1094 (808) | 723 (768) | 1423 (1014) | 1230 (1914)

6. Secondary Outcome: Pharmacokinetics (PK) (Assessed by Sampling and Testing for Drug and Metabolite Levels at Designated Time Points). Mean Terminal Elimination Half-life (t1/2,Term).
Description: Ibrutinib and PCI-45227 concentrations were measurable following once-daily dosing of ibrutinib in subjects with MM. The following time-points were included: 0hr, 1hr, 2hr, 7hr, 24hr post-dose. Ibrutinib terminal elimination half-life associated with the terminal slope (λz) of the semi-logarithmic plasma concentration-time curve, calculated as 0.693/λz on Day 8.
Time Frame: Procedure was performed up to 60 weeks.
Population: All subjects who received at least one dose of study treatment and had evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 13 | 16 | 18 | 43
hours | 7.76 (1.39) | 6.95 (0.821) | 8.42 (2.85) | 6.90 (1.81)

7. Secondary Outcome: Pharmacokinetics (PK) (Assessed by Sampling and Testing for Drug and Metabolite Levels at Designated Time Points). Mean Accumulation Ratio for AUC0-24h (Acc. Ratio AUC0-24h)
Description: Ibrutinib and PCI-45227 concentrations were measurable following once-daily dosing of ibrutinib in subjects with MM. The following time-points were included: 0hr, 1hr, 2hr, 7hr, 24hr post-dose. Acc. Ratio calculated as Day 8 ibrutinib AUC0-24h/ Day 1 ibrutinib AUC0-24h.
Time Frame: Procedure was performed up to 60 weeks.
Population: All subjects who received at least one dose of study treatment and had evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 13 | 16 | 18 | 43
Ratio | 2.75 (3.36) | 1.90 (1.64) | 1.88 (1.41) | 1.31 (0.830)

8. Secondary Outcome: Pharmacokinetics (PK) (Assessed by Sampling and Testing for Drug and Metabolite Levels at Designated Time Points). Mean Metabolite-to-Parent Ratio for Cmax (M/P Cmax)
Description: Ibrutinib and PCI-45227 concentrations were measurable following once-daily dosing of ibrutinib in subjects with MM. The following time-points were included: 0hr, 1hr, 2hr, 7hr, 24hr post-dose. Calculated as (PCI-45227 Cmax/PCI-45227 molecular weight)/(ibrutinib Cmax/ibrutinib molecular weight) on Day 8.
Time Frame: Procedure was performed up to 60 weeks.
Population: All subjects who received at least one dose of study treatment and had evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 13 | 16 | 18 | 43
Ratio | 0.952 (0.464) | 1.47 (0.632) | 1.39 (1.36) | 1.39 (0.746)

9. Secondary Outcome: Pharmacokinetics (PK) (Assessed by Sampling and Testing for Drug and Metabolite Levels at Designated Time Points). Mean Metabolite-to-Parent Ratio for AUC0-24h (M/P AUC0-24h)
Description: Ibrutinib and PCI-45227 concentrations were measurable following once-daily dosing of ibrutinib in subjects with MM. The following time-points were included: 0hr, 1hr, 2hr, 7hr, 24hr post-dose. Calculated as (PCI-45227 AUC0-24h/PCI-45227 molecular weight)/(ibrutinib AUC0-24h/ibrutinib molecular weight) on Day 8.
Time Frame: Procedure was performed up to 60 weeks.
Population: All subjects who received at least one dose of study treatment and had evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 13 | 16 | 18 | 43
Ratio | 1.44 (0.567) | 2.21 (0.985) | 1.90 (1.35) | 1.96 (0.923)

10. Secondary Outcome: Duration of Clinical Benefit Response (DCB)
Description: DCB is defined as the time from first observation of response to the time of disease progression.
Time Frame: From the date of first study treatment until disease progression per IMWG, up to 60 months
Population: Clinical benefit responders.
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 1 | 1 | 0 | 12
Months | 27.6 [27.6 to 27.6] | 3.7 [3.7 to 3.7] |  | 11.5 [2.8 to 46.3]

11. Secondary Outcome: Duration of Response (DOR)
Description: The time interval between the date of initial documentation of a response and the date of first documented evidence of progressive disease, death, or date of censoring for the subjects not progressed/died. The censoring date is the last adequate tumor assessment date.
Time Frame: up to 3 Years
Population: Responders
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | PCI-32765 420 mg Per Day | PCI-32765 560 mg Per Day, 40 mg Dexamethasone | PCI-32765 840 mg Per Day | PCI-32765 840 mg Per Day, 40 mg Dexamethasone
Number analyzed (Participants) | 0 | 1 | 0 | 2
Month |  | 3.7 [3.7 to 3.7] |  | 15.4 [3.6 to 27.2]

ADVERSE EVENTS:
Time Frame: Five Years
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 2/13 | 1/18 | 1/18 | 1/43
Serious Adverse Events (participants affected / at risk) | 6/13 | 6/18 | 7/18 | 12/43
Other Adverse Events (participants affected / at risk) | 12/13 | 18/18 | 17/18 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=13) | Cohort 2 (N=18) | Cohort 3 (N=18) | Cohort 4 (N=43)
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 4
Clostridium difficile infection (Infections and infestations) | 1 | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Aspergillus Infection (Infections and infestations) | 1 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Bacterial Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Bone Lesion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bronchopulmonary Aspergillosis (Infections and infestations) | 0 | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 0 | 0 | 1
Device Related Infection (Infections and infestations) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Epiglottitis (Infections and infestations) | 0 | 0 | 0 | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0
Hernia Pain (General disorders) | 0 | 1 | 0 | 0
Herpes Zoster Disseminated (Infections and infestations) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Lipase Increased (Investigations) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small Intestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Streptococcal Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Urinary tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Wound Secretion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=13) | Cohort 2 (N=18) | Cohort 3 (N=18) | Cohort 4 (N=43)
Diarrhoea (Gastrointestinal disorders) | 5 | 8 | 10 | 26
Fatigue (General disorders) | 3 | 7 | 9 | 21
Nausea (Gastrointestinal disorders) | 6 | 5 | 7 | 11
Anemia (Blood and lymphatic system disorders) | 4 | 6 | 6 | 12
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 | 6 | 3 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 5 | 4 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 2 | 12
Insomnia (Psychiatric disorders) | 1 | 5 | 1 | 13
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 2 | 7 | 8
Dizziness (Nervous system disorders) | 2 | 4 | 2 | 10
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 5 | 0 | 11
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 3 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 2 | 6
Pyrexia (General disorders) | 4 | 1 | 3 | 7
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 4 | 2 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 7
Constipation (Gastrointestinal disorders) | 1 | 4 | 2 | 5
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 2 | 3 | 6
Headache (Nervous system disorders) | 2 | 2 | 4 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2 | 1 | 5
Oedema Peripheral (General disorders) | 1 | 2 | 3 | 5
Vomiting (Gastrointestinal disorders) | 2 | 1 | 4 | 4
Abdominal Pain (Gastrointestinal disorders) | 3 | 2 | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 2 | 7
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 4
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 4
Urinary Tract Infection (Infections and infestations) | 0 | 2 | 3 | 5
Asthenia (General disorders) | 0 | 2 | 1 | 5
Contusion (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 2
Hypotension (Vascular disorders) | 1 | 1 | 1 | 4
Vision Blurred (Eye disorders) | 1 | 1 | 2 | 4
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 5
Blood Creatinine Increased (Investigations) | 0 | 2 | 1 | 3
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 1 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 4
Malaise (General disorders) | 0 | 1 | 2 | 4
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 2
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 3
Abdominal Distension (Gastrointestinal disorders) | 0 | 2 | 0 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 0 | 0 | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 4
Localised Infection (Infections and infestations) | 0 | 1 | 2 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 1
Pain (General disorders) | 0 | 0 | 2 | 3
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 2 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 3
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 3
Sinusitis (Infections and infestations) | 1 | 1 | 1 | 2
Weight Decreased (Investigations) | 1 | 2 | 0 | 3
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0 | 1 | 2
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Bandaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 2 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 1 | 1
Ear Discomfort (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Ear Congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Tympanic membrane disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 0 | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 0 | 2 | 0
Abnormal sensation in eye (Eye disorders) | 1 | 0 | 0 | 0
Asthenopia (Eye disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0
Choroidal infarction (Eye disorders) | 1 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0
Eye Pruritus (Eye disorders) | 0 | 0 | 0 | 1
Eyelid disorder (Eye disorders) | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 1
Iritis (Eye disorders) | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1
Ophthalmoplegia (Eye disorders) | 0 | 0 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Uveitis (Eye disorders) | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Angina bullosa haemorrhagica (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lip blister (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oral Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oral mucosa erosion (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Parotid gland enlargement (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tongue eruption (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tooth loss (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 3
Peripheral swelling (General disorders) | 1 | 0 | 2 | 1
Chest pain (General disorders) | 1 | 0 | 1 | 1
Feeling jittery (General disorders) | 2 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 1
Feeling abnormal (General disorders) | 1 | 0 | 0 | 1
Injection site bruising (General disorders) | 0 | 1 | 0 | 1
Crepitations (General disorders) | 1 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 1
Hernia pain (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 1
Unevaluable event (General disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 4
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Food allergy (Immune system disorders) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 1 | 1 | 1
Oral candidiasis (Infections and infestations) | 0 | 1 | 1 | 2
Paronychia (Infections and infestations) | 0 | 0 | 0 | 4
Ear Infection (Infections and infestations) | 0 | 0 | 1 | 2
Herpes Zoster (Infections and infestations) | 1 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 2
Candida infection (Infections and infestations) | 0 | 1 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 1 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 2
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 2
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Ear infection staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 1 | 0
Epiglottitis (Infections and infestations) | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Helicobacter infection (Infections and infestations) | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1
Measles (Infections and infestations) | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Systemic candida (Infections and infestations) | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 5
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Dental restoration failure (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Testicular injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0 | 0
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 2
Blood alkaline phosphatase decreased (Investigations) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0
Blood chloride increased (Investigations) | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1
Body temperature increased (Investigations) | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 1 | 0
Heart rate irregular (Investigations) | 0 | 0 | 0 | 1
Lymphocyte count increased (Investigations) | 1 | 0 | 0 | 0
Medical observation abnormal (Investigations) | 0 | 1 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 1
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 4 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle oedema (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 3
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 3
Syncope (Nervous system disorders) | 1 | 1 | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 0 | 2
Tremor (Nervous system disorders) | 0 | 0 | 0 | 2
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 1 | 0 | 0
Drooling (Nervous system disorders) | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0
Migraine with aura (Nervous system disorders) | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 3
Confusional state (Psychiatric disorders) | 1 | 1 | 0 | 1
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 3
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0
Affect lability (Psychiatric disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1
Claustrophobia (Psychiatric disorders) | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 2
Renal impairment (Renal and urinary disorders) | 0 | 1 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Breast ulceration (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Uterine cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Nail growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin warm (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1 | 2
Flushing (Vascular disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-04-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT01478581/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT01478581/SAP_001.pdf